CLINICAL TRIAL: NCT02957292
Title: A Randomized Controlled Trial to Compare the Menstrual Bleeding Profile Among Copper and 13,5mg Levonorgestrel-releasing IUD Users.
Brief Title: A Study to Compare the Menstrual Bleeding Profile Among Jaydess® and Copper Intrauterine Device (IUD) Users. COLIBRI STUDY (Copper and Levonorgestrel IUD Barcelona Research Initiative).
Acronym: COLIBRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-DIU-2015-85
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel; Intrauterine Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levonorgestrel IUD (Experimental): 13,5 mg Levonorgestrel intrauterine device
  Interventions: Drug: Levonorgestrel (13,5 mg) intrauterine device
- Copper IUD (Active Comparator): Copper (380mm2) intrauterine device
  Interventions: Device: Cooper (380mm2) intrauterine device

INTERVENTIONS:
Drug: Levonorgestrel (13,5 mg) intrauterine device
  Arms: Levonorgestrel IUD
Device: Cooper (380mm2) intrauterine device
  Arms: Copper IUD

SUMMARY:
The intrauterine device (IUD) is a long-term birth control method that has demonstrated high contraceptive efficacy and effectiveness due to its high compliance, adherence and persistence of use. The IUD has a global prevalence rate around 14% in women of reproductive age.

Side effects are the main reason for IUD use discontinuation. The most common reasons for copper IUD discontinuation are increased menstrual bleeding, irregular bleeding and dysmenorrhea, whereas in the case of 52mg Levonorgestrel IUD are irregular bleeding and amenorrhea.

In 2014, a new hormonal IUD containing13,5mg of Levonorgestrel was marketed in Spain. There are many studies comparing the two Levonorgestrel IUDs. However, there is any study comparing the IUD 13,5mg Levonorgestrel with classic copper IUDs.

The hypothesis of this trial is that Levonorgestrel (13,5mg) IUD users have a menstrual bleeding pattern with fewer days than Copper 380 mm2 IUD users.

This is a Phase IV, national single-center, randomized 1: 1, single-blind, comparative, parallel controled trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject.
* Parous or nulliparous women aged between 18 and 45 years who ask for an IUD as a contraceptive method.
* History of regular cyclic menstrual periods ranged from 21 to 35 days with non-excessive menstrual blood loss.

Exclusion Criteria:

* Absolute contraindications to IUD use, according to the World Health Organization Medical Eligibility Criteria.
* Contraindications to use 13,5 LNG-IUD.
* Anemia.
* Use of short or long-acting preparations containing sex hormones within the 12 weeks before the IUD insertion.
* Known bleeding irregularities.
* Pregnancy or breast-feeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Number of menstrual bleeding days | 90 days
  Daily recorded during 90 days treatment period
Amount of Menstrual bleeding | 90 days
  Classified using a 5-item Likert-like scale from none to heavy, a pictorial blood loss assessment chart (PBAC), and ferritin and haemoglobin blood test determinations

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain